CLINICAL TRIAL: NCT06696573
Title: Effectiveness of Proactive Versus On-Demand Pain Relief With Non-Steroidal Anti-Inflammatory Drugs During Medical Abortion at 13 to 22 Weeks at Hung Vuong Hospital
Brief Title: Effectiveness of Anti-Inflammatory Drugs for Preventing Pain Versus Treating Pain During Medical Abortion From 13 to 22 Weeks at Hung Vuong Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Le Thi Kieu Trang (Other)
Responsible Party: Sponsor-Investigator, Le Thi Kieu Trang, Doctor, Hung Vuong Hospital
Organization: Hung Vuong Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hung Vuong Hospital
Record Dates: First submitted 2024-11-09; First posted 2024-11-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pain Management; Anti-Inflammatory Agents, Non-Steroidal; Abortion, Spontaneous
MeSH Terms: conditions — Agnosia; Abortion, Spontaneous

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two arms: one group receiving prophylactic NSAIDs before the onset of pain during medical abortion and another group receiving NSAIDs on-demand. The study aims to compare the efficacy, safety, and overall pain management outcomes of the two strategies.
Masking Description: This is not applicable as this study is open-label, meaning both participants and care providers are aware of the intervention assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic NSAID Group for Pain Management in Medical Abortion (Experimental): Participants in this group will receive a prophylactic administration of a non-steroidal anti-inflammatory drug (NSAID) to manage pain before its onset during the medical abortion process for pregnancies between 13 and 22 weeks. The intervention will involve the use of a generic NSAID (e.g., Ibuprofen), administered in oral tablet form at a specified dosage, such as 400 mg. The medication will be taken prior to the expected onset of uterine contractions and will be monitored for efficacy and safety throughout the duration of the procedure. The administration may be repeated based on the clinical protocol, with an appropriate frequency adjusted according to the needs and response of the participant. The aim is to evaluate pain reduction, overall satisfaction, and any potential side effects or adverse events associated with this prophylactic approach.
  Interventions: Drug: Prophylactic NSAID Administration
- On-Demand NSAID Group for Pain Management in Medical Abortion (Experimental): Participants in this group will receive non-steroidal anti-inflammatory drugs (NSAIDs) on an as-needed basis during the medical abortion process for pregnancies between 13 and 22 weeks. The administration will occur once participants report experiencing pain, with the goal of managing pain symptoms as they arise. The intervention involves a specified dosage of a generic NSAID (e.g., Ibuprofen) in oral tablet form, typically 400 mg, administered as required to control pain. The effectiveness of on-demand NSAID administration will be evaluated in terms of pain relief, safety, and participant satisfaction throughout the procedure.
  Interventions: Drug: On-Demand NSAID Administration

INTERVENTIONS:
Drug: Prophylactic NSAID Administration — Participants in this arm will receive a prophylactic dose of a non-steroidal anti-inflammatory drug (NSAID) prior to the onset of pain during medical abortion procedures for pregnancies between 13 and 22 weeks. The intervention aims to reduce pain intensity throughout the process. The NSAID administration involves a specific dosage and schedule, adhering to safety guidelines and monitored for potential side effects.
  Arms: Prophylactic NSAID Group for Pain Management in Medical Abortion
Drug: On-Demand NSAID Administration — Participants in this group will receive a non-steroidal anti-inflammatory drug (NSAID), such as Ibuprofen, in oral tablet form at a dose of 400 mg. The drug will be administered as needed when participants report experiencing pain during the medical abortion process for pregnancies between 13 and 22 weeks. The goal of this intervention is to provide pain relief in response to individual needs, with administration and dosage adjusted as clinically indicated. Monitoring will occur to assess the efficacy, safety, and patient response to the on-demand approach.
  Arms: On-Demand NSAID Group for Pain Management in Medical Abortion

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of non-steroidal anti-inflammatory drugs (NSAIDs) for prophylactic pain relief compared to on-demand pain relief during medical abortion for pregnancies between 13 and 22 weeks at Hung Vuong Hospital in Ho Chi Minh City. The main questions it aims to answer are:

1. Does prophylactic use of NSAIDs reduce pain compared to on-demand use during medical abortion?
2. What are the potential adverse effects of NSAIDs in this context?

Researchers will compare a group receiving prophylactic NSAIDs to a control group receiving on-demand pain relief to determine if the prophylactic approach leads to improved pain management outcomes.

Participants will:

* Be given NSAIDs either as a preventative measure or upon the onset of pain.
* Be monitored for pain levels using validated pain scales, any side effects, and outcomes of the abortion procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years or older.
* No mental illness.
* Gestational age between 13 and 22 weeks (based on the last menstrual period with a regular menstrual cycle and accurate recall of the last menstrual period, or based on a first-trimester ultrasound) with an indication of stillbirth, fetal malformation requiring termination, or voluntary abortion with counseling and understanding of the abortion procedure.
* Willing to participate in the study.
* Capable of reading and signing the informed consent form.
* Able to provide personal information independently.

Exclusion Criteria:

* Medical conditions contraindicating medical abortion: bleeding disorders, anticoagulant use, moderate to severe anemia.
* Cardiovascular conditions: heart failure, mitral valve stenosis, embolism, uncontrolled hypertension.
* Other medical conditions: renal failure, adrenal gland disorders, severe asthma, liver and biliary diseases, glaucoma.
* Active pelvic inflammatory disease or acute genital infections.
* Previous uterine surgery.
* Placenta previa or central placenta previa.
* Uterine malformations.
* History of allergy to NSAIDs, Mifepristone, or Misoprostol.
* Unwillingness to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparing the Effectiveness of Prophylactic NSAID Pain Relief Versus On-Demand Treatment in Cases of Medical Abortion Indicated for Gestational Age 13 to 22 Weeks at Hung Vuong Hospital | Data will be collected from the initiation of medical abortion treatment through abortion completed
  Change in pain scores measured using the Visual Analog Scale (VAS) in millimeters, assessed from baseline to the end of treatment during medical abortion procedures for gestational ages between 13 to 22 weeks. Pain levels will be recorded at regular intervals during and after the administration of prophylactic versus on-demand NSAID treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam